CLINICAL TRIAL: NCT04518631
Title: Effects of Mindfulness Training on Emotional Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Lam Shui-fong, Director of Jockey Club Peace and Awareness Mindfulness Culture in Schools Initiative, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UHongKong(PandA)
Record Dates: First submitted 2020-08-12; First posted 2020-08-19 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Mental Health Issue
Keywords: mindfulness; teacher mental health; emotional care; mindfulness-based intervention for teachers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8-week mindfulness program (Experimental): 8-week .b Foundations course
  Interventions: Behavioral: 8-week mindfulness program
- Wait-list control (No Intervention): Participants in wait-list control group will receive the same intervention, two months after their counterparts in experimental group completed the intervention.

INTERVENTIONS:
Behavioral: 8-week mindfulness program — The .b Foundations course is an 8-week mindfulness program developed by Mindfulness in Schools Project (MiSP) for school teachers and personnel. It includes a taster session and 8 weekly sessions. Each session lasts for 1.5 hours with a specific theme (e.g. Lesson 1 waking up from autopilot). Formal and informal mindfulness practices (e.g. mindful eating, body scan, mindful walking, habit releaser etc.), psychoeducation, cognitive exercises, inquiry, and home practice are involved.
  Arms: 8-week mindfulness program

SUMMARY:
Teachers in Hong Kong are susceptible to professional stress and its associated psychosomatic illnesses. To enhance teachers' well-being, mindfulness training is conducted in local schools. The present study is a randomized controlled trial to investigate 1) the effects of mindfulness training on teachers' well-being (i.e. general health, positive affect, life satisfaction, stress, negative affect), and 2) the mechanisms underlying the effectiveness of mindfulness (i.e. emotional care strategies including anchoring, decentering, and acceptance). Participants will be randomized to either intervention (8-week .b Foundations/ .begin course) or waiting-list control condition. They will complete survey before (baseline), after (post-intervention), and two-months (follow-up) after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or above
* Working in local schools or education institutions
* Willing to participate in mindfulness training voluntarily

Exclusion Criteria:

* Experiencing severe or unstable mental health condition currently
* Completed 8-week mindfulness training previously
* Unwilling to go by random assignment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in General Health | Baseline, Immediately after intervention, Two-months after intervention
  General Health Questionnaire (GHQ), 12 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Stress | Baseline, Immediately after intervention, Two-months after intervention
  Perceived Stress Scale (PSS), 10 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Anchoring | Baseline, Immediately after intervention, Two-months after intervention
  5 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Decentering | Baseline, Immediately after intervention, Two-months after intervention
  Non Reactivity Subscale of Chinese Five Facet Mindfulness Questionnaire (FFMQ-C), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Acceptance | Baseline, Immediately after intervention, Two-months after intervention
  Acceptance subscale of Cognitive and Affective Mindfulness Scale-Revised (CAMS-R), 3 items, 5-point Likert scale ranging from 1 (never) to 5 (always)

SECONDARY OUTCOMES:
Change in Life satisfaction | Baseline, Immediately after intervention, Two-months after intervention
  Life Satisfaction Questionnaire, 5 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Positive affect | Baseline, Immediately after intervention, Two-months after intervention
  Positive and Negative Affect Schedule (PANAS), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Negative affect | Baseline, Immediately after intervention, Two-months after intervention
  Positive and Negative Affect Schedule (PANAS), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Reappraisal | Baseline, Immediately after intervention, Two-months after intervention
  Reappraisal subscale of Emotion Regulation Questionnaire (ERQ), 6 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Suppression | Baseline, Immediately after intervention, Two-months after intervention
  Suppression subscale of Emotion Regulation Questionnaire (ERQ), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Distraction | Baseline, Immediately after intervention, Two-months after intervention
  5 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Mindfulness | Baseline, Immediately after intervention, Two-months after intervention
  Cognitive and Affective Mindfulness Scale-Revised (CAMS-R), 12 items, 5-point Likert scale ranging from 1 (never) to 5 (always)

CONTACTS AND LOCATIONS:
Locations (1):
- Jockey Club "Peace and Awareness" Mindfulness Culture in Schools Initiative, Faculty of Social Sciences, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided